CLINICAL TRIAL: NCT00123500
Title: ACTION! Wellness Program for Elementary School Personnel
Brief Title: Wellness Program for Elementary School Personnel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University School of Public Health and Tropical Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Larry S. Webber, Professor, Tulane University School of Public Health and Tropical Medicine
Organization: Tulane University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 234; R01HL079509 (NIH); NCT00122967 (obsolete NCT alias)
Record Dates: First submitted 2005-07-21; First posted 2005-07-25 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Obesity; Cardiovascular Diseases
MeSH Terms: conditions — Obesity; Cardiovascular Diseases | interventions — Diet; Exercise; Environment; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Worksite Intervention
  Interventions: Behavioral: Diet; Behavioral: Physical Activity; Behavioral: Environment
- 2 (Placebo Comparator): Control Group
  Interventions: Other: Control Group

INTERVENTIONS:
Behavioral: Diet — Diet
  Arms: 1
Behavioral: Physical Activity — Physical Activity
  Arms: 1
Behavioral: Environment — Environment
  Arms: 1
Other: Control Group — Control Group
  Arms: 2

SUMMARY:
The goal of the project is to develop, implement, and evaluate, through a randomized controlled trial at a worksite, an intervention to promote increased physical activity behavior and healthier eating behavior to reduce overweight and obesity among elementary school personnel.

DETAILED DESCRIPTION:
BACKGROUND:

The dramatic increase in the prevalence of overweight and obesity among adults in the United States during the past two decades is related to increased cardiovascular disease, hypertension, dyslipidemia, diabetes, and other chronic diseases. With 63.9% of working-age adults employed, worksites are targets for prevention and intervention programs to control overweight and obesity. Worksite interventions have the potential to reach a large number of individuals in a common and shared environment.

DESIGN NARRATIVE:

This is a group-randomized trial involving 20 elementary schools in Jefferson Parish public schools. Schools will be the unit of randomization; 10 schools will be randomly allocated to implement the intervention, and 10 schools will serve as controls. The primary aim of the program is to reduce mean body weight. Secondary aims relate to changes at both the individual level and the environmental level. The intervention will address the two major determinants of overweight and obesity: physical activity and diet. A School Wellness Committee at each site will be instrumental in identifying and implementing components of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults with no contraindications to participating in an intervention to improve eating and exercise behaviors
* Healthy adults with no contraindications to participating in any of the measurement procedures

Exclusion Criteria:

* Inability to participate in routine physical activity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1202 (Actual)
Dates: Start 2004-09; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Body mass index (BMI) | Measured at the end of the second year of intervention

SECONDARY OUTCOMES:
24-hour dietary recall | Measured at baseline (Fall 2006) and follow-up (Fall 2008)

CONTACTS AND LOCATIONS:
Overall Officials: Larry Webber, PhD, Principal Investigator — Tulane University
Locations (1):
- Tulane University, New Orleans, Louisiana, United States